CLINICAL TRIAL: NCT03487835
Title: Role of Kinesiology Tape in Reducing Physiological Fall Risk in Older Adults
Brief Title: Role of Kinesiology Tape in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/298
Record Dates: First submitted 2017-11-15; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2017-11

CONDITIONS: Older Adult
Keywords: Athletic tape. Accidental Falls. Aging.
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape group (Experimental)
  Interventions: Other: Kinesiotape
- Control group (Experimental)
  Interventions: Other: No application

INTERVENTIONS:
Other: Kinesiotape
  Arms: Kinesiotape group
Other: No application — This group have no application during study time
  Arms: Control group

SUMMARY:
Aim: The present study aimed to investigate the role of Kinesiology ('Kinesio') tape in the physiological risk of falling in older adults.

Methods: Twenty two older adults aged over 65 years and living in nursing homes. After assessment of demographic information, they were randomized into one of two groups [(Kinesio tape (n = 22) and control (n = 20)]. Kinesio tape was applied on the Kinesio tape group only and worn during a 2-week intervention period. Participants were evaluated with the Visual Analog Scale, Berg Balance Scale, Timed Up and Go Test, Mini-Mental State Examination, 30-Second Sit to Stand test and Functional Independent Measurement instrument at baseline, after 2 weeks of application and at 2-week follow-up.

DETAILED DESCRIPTION:
Measures After participant demographics data (age, daily medication etc.) and their history of falls information been collected, the Berg Balance Scale (BBS), Functional Independence Measure (FIM), and Visual Analog Scale (VAS) were administered along with the Timed Up and Go test (TUG) and 30-Second Sit to Stand test (30s STS).

2.1. History of falls Participating adults were then asked about another resident's experience of falls in the preceding year. Interviews were conducted verbally.

2.2. The visual analog scale The VAS is a pain-intensity measurement scale that is both effective and simple to use; the reliability and validity of the VAS have been previously determined. To determine perceived body pain, individuals are asked to mark the intensity of their existing pain on a 10-cm scale where a range of numbers-from 0 (no pain) to 10 (unbearable pain)-are displayed to determine body pain (Tyler, Jensen, Engel and Schwartz, 2002).

2.3. The functional independence measure The FIM analyses two aspects of disability: motor and cognitive functions. The FIM is comprised of six functional categories: self-care, sphincter control, mobility, locomotion, communication, and social perception. A total of 18 activities are evaluated by the FIM to determine functional independence; a seven-point scale is used to evaluate each activity with the highest-possible score for the scale being 126 (Küçükdeveci, Yavuzer, Elhan, Sonel and Tennant, 2001).

2.4. The timed up and go The TUG test is an objective, reliable and simple measure aimed at evaluating balance and functional mobility; the TUG test can also be used to assess the risk of falling. Scores are calculated by measuring the number of seconds it takes for a participant to complete the test. The use of a walking aid is permitted during the test (Amold & Faulkner, 2007).

2.5. 30-Second sit to stand The 30s STS test measures leg strength; the test records the number of times a patient can go from a sitting to a standing position within a 30-secondperiod. For the safety of the participant, the chair used for the test should be rested against a wall to ensure that it does not slip. The patient's transformation from a standing into a sitting position should be performed in full (Whitney et al., 2005).

2.5. The berg balance scale The BBS assesses balance by testing a patient's ability to maintain their balance while performing functional activities. The Berg Balance Scale is comprised of 14 items; each section is graded on a scale from 0 (bad) to 4 (best). Higher scores indicate better balance. Scores of 0-20 signify high risk, those of 21-40 signify medium risk and those of 41-64 signify low risk (Bogle & Newton, 1996).

2.6. The mini-mental state examination The MMSE assesses an individuals' mental function. The standardization of this scale was established in Turkish by Güngen, Ertan, Eker, Yaşar, and Engin (2002); the scale is easily applicable and provides information regarding a participant's cognitive impairment. The highest possible score is 30, with higher scores indicating good cognitive status. Scores lower than 23-24 are generally suggestive of an 'abnormal' cognition; additional levels of score breakdown specified (Güngen, Ertan, Eker, Yaşar, Engin, 2002).

3. 'Kinesio' tape application The original 'Kinesio' tape (5cm wide) for this study. Only those participants in the 'Kinesio' tape group only were taped; tape was applied in accordance with Kenzo Kase's 'Kinesio' taping manual (Kase et al., 1996; Kase et al., 2003). Before application of the tape, the area of application was wiped with water containing 70% alcohol; anything that might prevent the tape from adhering to patient's skin eliminated prior to the application. The length of the extremity subject to the tape's application was measured and three I-shaped tapes were cut accordingly; one tape was applied to the ankle and the other two tapes were applied along the base of the extremity to support the arches of the foot, starting around the malleoli (Figure 2 and 3).

Consequently, the patient's ankle and foot arches were supported; additionally, the researchers aimed to increase ankle stability and the proprioceptive sense the tape provided the foot and ankle. The application was performed by stretching the tape original length between 25-75%, according to the technique outlined by Kase, Wallis, and Kase (2003). An expert physiotherapist with a 'Kinesio' tape certificate applied the tape while the participant was in a sitting position, and was also responsible for taking all the appropriate measurements.. Individuals in the 'Kinesio' group were visited every other day for two-week intervention period. Tapes were verified during this period, and those with deformities were removed and new ones were applied instead. All participants had their tape removed and reapplied every three days. All participants lived in nursing homes and their nursing-home staff were informed about the study protocol. In particular, participants were informed that the tape did not need to be removed during bathing or situations such as getting dressed. After the two-week intervention period, the TUG, the BBS, 30s STS, FIM and VAS were re-administered to both the 'Kinesio' tape group and the control. During the two weeks that followed the second measurement, no 'Kinesio' tape application was conducted on either group. Two weeks following the end of the intervention period, a third set of measurements were taken from each group. In summary, three measurements were administered to each group, these included: one at baseline, prior to 'Kinesio' taping application; 1st measurement; one following application, 2nd measurement; and one after a two-week follow-up period, 3rd measurement. After study had been completed, the 'Kinesio' tape application was offered to individuals in the control group if they desired.

ELIGIBILITY:
Inclusion Criteria:

* After signing the consent form, individuals who agreed to participate underwent the Timed Up and Go test. Participants whose the Timed Up and Go (TUG) test score was over 13 s (Fig. 1),14) who showed full cooperation and who had no hearing or vision problems that would affect the ability to participate in the study evaluation methods were included in the study

Exclusion Criteria:

* Bedridden older adults, those with an acute disease or infection, those with cognitive problems [assessed by the Mini-Mental State Examination (MMSE)], a lower extremity orthosis or prosthesis, neurological issues and those who had endured a break in their lower extremities within the last 3 months were excluded from the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test and Berg Balance Scale | 4 days/ two weeks
  the application of 'Kinesio' tape has positive effects on functional mobility and balance in older adults
the effect of time | follow up two weeks
  The effects of 'Kinesio' tape last for at least two weeks after application

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi YK, Nam CW, Lee JH, Park YH. The Effects of Taping Prior to PNF Treatment on Lower Extremity Proprioception of Hemiplegic Patients. J Phys Ther Sci. 2013 Sep;25(9):1119-22. doi: 10.1589/jpts.25.1119. Epub 2013 Oct 20. PMID 24259927
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Result] Hawk C, Hyland JK, Rupert R, Colonvega M, Hall S. Assessment of balance and risk for falls in a sample of community-dwelling adults aged 65 and older. Chiropr Osteopat. 2006 Jan 27;14:3. doi: 10.1186/1746-1340-14-3. PMID 16441893